CLINICAL TRIAL: NCT06296680
Title: The Effect of Reiki Applied to Cancer Patients on Pain, Anxiety, and Stress Levels: A Randomized Controlled Study
Brief Title: Reiki for Cancer: Pain, Anxiety, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sevcan Oz Kahveci, Research Assistant, Ege University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: EGE_UNI_SEVCAN_OZ_KAHVECI_0001
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Therapeutic Touch; Cancer
Keywords: Reiki; Cancer; Pain; Anxiety; Stress; Nursing
MeSH Terms: conditions — Neoplasms; Pain; Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study is a three-arm intervention trial. Reiki was applied to the intervention group, Sham Reiki to the placebo group, and Progressive Relaxation Exercise to the control group. The effects of these three methods applied to cancer patients on their levels of pain, anxiety, and cortisol were examined.
Who Masked: Participant, Investigator
Masking Description: In order to prevent assessment bias, blinding was implemented throughout the collection of data from patients, evaluation of the effectiveness and reliability of the applied dependent variables, data processing, reporting, and statistical analysis. The researcher was provided with a randomization list by a statistical expert. The researcher was included in the study without knowing which group the patients would be assigned to, and the patients were also enrolled without knowledge of their group assignment. Therefore, this study was conducted as a three-arm, double-blind, randomized follow-up study in the experimental research model, with intervention, placebo, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): In the intervention group, patients received an energy therapy called Reiki. Reiki was administered to cancer patients for four consecutive days at specified times. During this procedure, while the patient was in the supine position, the researcher's hands were placed approximately two to three centimeters above the chakra regions of the patient, covering the seven chakra areas as well as the areas experiencing pain. The application lasted a total of 25-30 minutes. Silence was maintained in the patient's room during the intervention.
  Interventions: Other: Reiki
- Sham Reiki (Sham Comparator): In the placebo group, patients received Sham Reiki. Sham Reiki was administered to cancer patients for four consecutive days at specified times. During this procedure, while the patient was in the supine position, Sham Reiki practitioner's hands were placed approximately two to three centimeters above the chakra regions of the patient, covering the seven chakra areas as well as the areas experiencing pain. The application lasted a total of 25-30 minutes. Silence was maintained in the patient's room during the intervention.
  Interventions: Other: Sham Reiki
- Progressive Relaxation Exercise (Active Comparator): Silence was maintained in the patient's room during the intervention. At the beginning of the session, the patient is asked to assume the most comfortable seated or supine position. Then, they are instructed to close their eyes, take deep breaths, direct their thoughts to their own body and the muscle groups being treated, notice the tension and relaxation in the muscle groups during the exercise, and continue to breathe regularly. This practice was conducted in four parts of the body: hands and arms; face and shoulders; chest, abdomen, hips; legs and feet.
  Interventions: Other: Progressive Relaxation Exercise

INTERVENTIONS:
Other: Reiki — The patients in the intervention group received Reiki to the seven chakra regions and additional areas with pain for a total duration of 25-30 minutes for four consecutive days. On the 4th day, pain and anxiety levels of the patients were evaluated after the last applications. On the 21st day, pain and anxiety levels were evaluated, State Anxiety Scale and Perceived Stress Scale were administered, and serum cortisol level was evaluated in the morning before the start of chemotherapy. At the 3rd month follow-up, pain and anxiety levels, state anxiety scale and perceived stress scale were evaluated.
  Arms: Reiki
Other: Sham Reiki — The patients in the placebo group received Sham Reiki to the seven chakra regions for a total duration of 25-30 minutes for four consecutive days. On the 4th day, pain and anxiety levels of the patients were evaluated after the last applications. On the 21st day, pain and anxiety levels were evaluated, State Anxiety Scale and Perceived Stress Scale were administered, and serum cortisol level was evaluated in the morning before the start of chemotherapy. At the 3rd month follow-up, pain and anxiety levels, state anxiety scale and perceived stress scale were evaluated.
  Arms: Sham Reiki
Other: Progressive Relaxation Exercise — PRE group patients received PRE for four consecutive days. On the 4th day, pain and anxiety levels of the patients were evaluated after the last applications. On the 21st day, pain and anxiety levels were evaluated, State Anxiety Scale and Perceived Stress Scale were administered, and serum cortisol level was evaluated in the morning before the start of chemotherapy. At the 3rd month follow-up, pain and anxiety levels, state anxiety scale and perceived stress scale were evaluated.
  Other Names: the patients in the control group received Progressive Relaxation Exercise.
  Arms: Progressive Relaxation Exercise

SUMMARY:
The goal of this clinical trial is to investigate the effects of Reiki, Sham Reiki, and Progressive Relaxation Exercise on the levels of pain, anxiety, and stress in cancer patients.

The main questions it aims to answer are:

* Question 1: The effect of Reiki applied to cancer patients on the level of pain within the time series is higher in favor of the intervention group.
* Question 2: The effect of Reiki applied to cancer patients on the level of anxiety within the time series is higher in favor of the intervention group.
* Question 3: The effect of Reiki applied to cancer patients on cortisol levels within the time series is higher in favor of the intervention group.
* Question 4: The effect of Reiki applied to cancer patients on the level of stress within the time series is higher in favor of the intervention group.
* Participants have answered the questions in the Individual Identification Form, Visual Comparison Scale, State Anxiety Scale and Perceived Stress Scale and serum cortisol levels were evaluated in the pretest.
* Afterwards, the patients in the intervention group received Reiki for four consecutive days, the patients in the placebo group received Sham Reiki, and the patients in the control group received Progressive Relaxation Exercise.
* The patients in the experimental group received Reiki to the seven chakra regions and additional areas with pain for a total duration of 25-30 minutes for four days, with an average of three minutes.
* The patients in the placebo group received Sham Reiki to the seven chakra regions for a total duration of 25-30 minutes for four days, with an average of three minutes.
* Progressive Relaxation Exercise (PRE) group patients received PRE for four days.
* On the 4th day, pain and anxiety levels (0-10 Likert-type scale) of the patients were evaluated after the last applications.
* On the 21st day, the day of the next chemotherapy cycle, pain and anxiety levels were evaluated, state anxiety scale and perceived stress scale were administered, and serum cortisol level was evaluated in the morning before the start of chemotherapy.
* At the 3rd month follow-up, pain and anxiety levels (0-10 Likert-type scale), state anxiety scale and perceived stress scale were evaluated.

DETAILED DESCRIPTION:
Patients were assigned to intervention, placebo, and control groups according to a randomization list. Laboratory fees for serum cortisol analyses were covered from a separate budget to ensure patients under the coverage of the Social Security Institution did not experience any deduction of fees. For each patient consenting to participate in the study, contact was made with the Ege University Faculty of Medicine Project and Special Services Coordination Center (PROKOM) for "Research Patient Identification", followed by contacting the Hospital Information Processing Department to open a "Research Patient" record. Laboratory requisitions for patients were made by the attending physician. Following serum cortisol analyses, data from the "Individual Identification Form, Visual Analog Scale, State Anxiety Inventory, Perceived Stress Scale" were collected from patients. Patients consenting to participate in the study were then initiated on treatment plans by a researcher with Level One certification in Reiki and PGE (Progressive Relaxation Exercise). Sham Reiki was administered by Sham Reiki practitioners. Patient rooms in the clinic were single occupancy, and efforts were made to control noise during interventions. Any accompanying family member/caregiver present in the room during the intervention was asked to leave for the duration of the application.

* Intervention Group (Reiki Group):
* Pre-test: Prior to initiating Reiki application, blood samples were obtained from the patients to assess serum cortisol levels; subsequently, data from the "Individual Identification Form, Visual Analog Scale, State Anxiety Inventory, Perceived Stress Scale" were collected by the researcher through face-to-face interviews. Reiki was administered for four days at designated times. Reiki was applied for a total duration of 25-30 minutes, with approximately three minutes per chakra region and the area of pain, while the patient was in a supine position, and the researcher's hands were positioned two to three centimeters above the chakra regions.
* Fourth-day follow-up: Data from the Visual Analog Scale were collected, and anxiety scores were evaluated.
* Twenty-first-day follow-up: Patients' serum cortisol levels were re-evaluated just before the start of their next chemotherapy session (between days 21-28), before initiating their current medical treatment (patients use cortisol alongside chemotherapy treatment), and data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected.
* Three-month follow-up: Data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected from the patients.
* Placebo Group (Sham Reiki Group):
* Pre-test: Prior to initiating Sham Reiki application, blood samples were obtained from the patients to assess cortisol levels; subsequently, data from the "Individual Identification Form, Visual Analog Scale, State Anxiety Inventory, Perceived Stress Scale" were collected by the researcher through face-to-face interviews. Sham Reiki was administered for four days at designated times. In this study, Sham Reiki practitioners mimicked a Reiki session by moving their hands over the patient's body in a specific sequence for a duration of 25-30 minutes. Sham Reiki was applied for a total duration of 25-30 minutes, with approximately three minutes per chakra region and the area of pain, while the patient was in a supine position, and the practitioner's hands were positioned two to three centimeters above the chakra regions. Sham Reiki practitioners consisted of nurses who did not believe in the transfer of biological field energy.
* Fourth-day follow-up: Data from the Visual Analog Scale were collected, and anxiety scores were evaluated.
* Twenty-first-day follow-up: Patients' serum cortisol levels were re-evaluated just before the start of their next chemotherapy session (between days 21-28), before initiating their current medical treatment, and data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected.
* Three-month follow-up: Data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected from the patients.
* Control Group (PGE Group):
* Pre-test: Prior to initiating PGE application, blood samples were obtained from the patients to assess cortisol levels; subsequently, data from the "Individual Identification Form, Visual Analog Scale, State Anxiety Inventory, Perceived Stress Scale" were collected by the researcher through face-to-face interviews. Patients received PGE for four days.
* Fourth-day follow-up: Data from the Visual Analog Scale were collected again, and anxiety scores were evaluated.
* Twenty-first-day follow-up: Patients' serum cortisol levels were re-evaluated just before the start of their next chemotherapy session (between days 21-28), before initiating their current medical treatment, and data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected again.
* Three-month follow-up: Data from the Visual Analog Scale, State Anxiety Inventory, and Perceived Stress Scale were collected from the patients.

ELIGIBILITY:
Inclusion Criteria:

* Conscious
* Aged 18 and over
* Without serious mental disorders (Bipolar Disorder, Schizophrenia, Schizoaffective Disorder, Major Depression, Personality Disorders)
* Without visual and hearing impairments
* Capable of verbal communication
* Never received Reiki before
* Patients scoring 36 or above on the Perceived Stress Scale were included in the study.

Exclusion Criteria:

Patients using cortisol were not included in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Stress levels | In the pre-test and on the 21st-day follow-up
  Stress levels of the patients was measured by Perceived Stress Scale and serum cortisol levels. The 14-item five-point Likert-type scale consists of two factors. The lowest score a participant can obtain from this scale is 0 and the highest score is 56. A high score indicates that the person's perception of stress is high. A high total score means that the perceived stress level is high. As a result of the score between 0-35, it can be said that the participants are in a positive stress level, they can cope with stress effectively and the coping mechanisms they use are functional. It can be said that the methods used by the participants with a score range between 36-56 are not functional, that is, they cannot cope with stress effectively. Prior to initiating the interventions, blood samples were obtained from the patients to assess serum cortisol levels; on the twenty-first day follow-up, they were reassessed before the commencement of medical treatment.

SECONDARY OUTCOMES:
Anxiety levels | In the pre-test, on the 4th-day, on the 21st-day and 3rd month
  Anxiety level of the patients was evaluated with 0-10 Likert-type scale and State Anxiety Inventory (STAI-S). Anxiety level of the patients was evaluated with 0-10 Likert-type scale and State Anxiety Inventory (STAI-S). The original form was designed by Spielberger et al. (1970) to determine the state and trait anxiety levels of individuals separately. The scale can be administered to individuals aged 14 years and older. There are 20 items in the scale and the scale provides information about the anxiety level of the patient. There are ten inverted statements in the scale
Pain levels | In the pre-test, on the 4th-day, on the 21st-day and 3rd month
  The pain level of the patients was evaluated with a 0-10 Likert-type scale called Visual Analogue Scale (VAS). The VAS is a scale used to determine the level of pain between "0: no pain" and "10: unbearable pain". VAS is considered a reliable and valid measurement tool in repeated measurements. It is used to assess the severity of acute pain. It has been noted to have higher sensitivity compared to other methods in evaluating pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)